CLINICAL TRIAL: NCT03961750
Title: TAIC - Implementation of Student-led Otago Classes for a Falls Risk, Community Dwelling Older Adult Population
Brief Title: TAIC: Student-led Exercise for Older Adults at Risk of Falling
Acronym: TAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAIC
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Falls; Exercise
Keywords: Older Adult; OTAGO; Student led
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Pre Post test single cohort feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A feasibility study examining a single patient group undertaking a 12 week, student-led, OTAGO exercise class for community dwelling older adults at Glasgow Caledonian University. OTAGO consists of progressive strength and balance exercises.
  Interventions: Other: OTAGO

INTERVENTIONS:
Other: OTAGO — 12 Week exercise class programme
  Other Names: Otago exercise classes

SUMMARY:
The National Records of Scotland population projections show the pension age population increasing by 25% over the next 25 years. Falls are a major cause of hospitalisation in older adults, one in three community dwelling older adults over 65 years of age fall each year. There is a need to explore novel methods of delivering care to a growing older adult population. A programme of exercise called OTAGO has been found to reduce the number of falls for older adults. Several studies have explored the use of students to lead exercise interventions but these have not included assessing the impact to student educational experiences and outcomes with varying degrees of success on patient outcomes and no adverse events.

Research Aim: To examine the feasibility of a student-led exercise intervention in improving falls risk outcomes for community dwelling older adults at risk of falling referred from NHS falls services.

Study Design: A feasibility study examining a single patient group undertaking a 12 week, student-led, OTAGO exercise class for community dwelling older adults at Glasgow Caledonian University. OTAGO consists of progressive strength and balance exercises.

Participants will be screened, invited to consent to the trial, asked to undertake the 12 week intervention and assessed using physical measures before and after the trial and face to face interviews after the trial.

Recruitment will be through the NHS Greater Glasgow and Clyde and Lanarkshire community falls teams and the exercise delivery is consistent with usual care, the main difference is the location and student leaders. Students are qualified OTAGO Leaders.

Funding has been received from AGILE the Chartered Society of Physiotherapists professional network working with older adults.

Student educational experiences and outcomes will be assessed over the study period and are included in a separate study protocol

DETAILED DESCRIPTION:
In the TAIC study we will examine the feasibility of a student-led exercise intervention in improving falls risk outcomes for community dwelling older adults at risk of falling. Additionally, we will examine the impact on students education and learning from leading an exercise intervention for community dwelling older adults at risk of a fall. Although we aim to submit this aspect of the study as a separate protocol.

The aim will be explored concurrently using a pre-post test design.

Principal Aim:

To examine the feasibility of a student-led exercise intervention in improving falls risk outcomes for community dwelling older adults at risk of falling referred from NHS Falls services.

Design and Intervention:A pre-post test single cohort design of a 12 week OTAGO exercise intervention of 3 times a week, 60 minute exercise sessions through a combination of home exercises and 1-2 face to face classes per week, dependant on availability of students and participants.

Rationale: Feasibility or pilot study design can be used in physical activity related interventions to inform practice, to gain an understanding of resource requirements, to inform management and to advance scientific enquiry. A paper by Bowen (2009) further outlines feasibility study design in public health. Bowen (2009) outlines eight areas of focus that will be explored in this study; adaptability, demand, implementation, practicality, adaptation, integration, expansion and limited-efficacy testing. Feasibility studies can also suffer from poor methodological quality and El-Kotob (2018) have outlined a number of challenges to undertaking physical activity research using the PICO framework. The below methodology has been designed using these eight areas of focus and potential methodological flaws.

The feasibility of this intervention will be reviewed using mixed methods research. Quantitative review of feasibility will include using pre-post outcome measure assessments and analysis, referral rates of participants, student volunteer numbers and adherence rates for class and home exercises. Qualitatively we will conduct a survey of student confidence in managing community dwelling older adults at risk of falls; additionally both students and participants will undertake semi-structured interviews to examine in more depth their experience in this study.

Methodologically we will not be using a control group as the OTAGO programme is well established as an effective intervention for community dwelling older adults at risk of a fall and would be potentially harmful to their current care to withhold this intervention (Robertson and Campbell 2001, Public Health England, 2017, Royal College of Physicians, 2012). Fidelity of treatment will be maintained by incorporating a break in the programme to allow students to complete their exams while still affording patients the full 12 week OTAGO intervention. The inclusion criteria will be the same as current care with only one major change that participants must not be cognitively impaired to ensure consent, for inclusion in the feasibility study, is clearly obtained and to ensure student volunteers can manage a group of individuals who can follow instructions safely.

Sampling:

Eligibility Criteria We will recruit approximately 15 participants to this study through direct referral from NHS falls services based in NHS GGC and NHS Lanarkshire. Participants will be identified by HCPC registered physiotherapists and support workers. Information leaflets will be provided to any potential participant by the NHS falls service team and a referral form will be completed.

Sampling Method: Convenience sampling will be used based on the eligible patients referred to the NHS falls services during the recruitment period. As this is a feasibility study aimed at gauging service demand and future implementation it is necessary to see the scope of referrals to gauge the potential for future classes. This method also ensures that no participants are disadvantaged by missing this evidence based intervention as any participants after saturation will simply be referred back to the NHS to another falls class in their area.

PARTICIPANT INVOLVEMENT

Outcome Measures and time points:

The TAIC study is due to start recruiting as soon as feasible but likely September 2019 with the classes starting at the end of October 2019 and lasting initially for 8 weeks until students have a christmas break and then re-starting in late January for four more weeks.

Outcome measure assessment will be undertaken approximately 1 week prior to attending the 1st OTAGO classes (Week -1) as part of the 12-week intervention (Week 1-12) and approximately 1 week after the final session (Week +1). Comparison of results will be difference between pre and post scores for this single cohort, Week -1 compared to Week +1.

Outcome measure assessments - student volunteers trained as OTAGO instructors and trained by the chief investigator in undertaking specific outcome measures. Outcome measure training will involve a 1-hour introduction to the outcome measures to be used and then an assessment session using health control volunteers over two separate days to ensure consistency of scoring and procedure. The chief investigator will facilitate this training.

Semi-structured interviews - Dr Fiona Kennedy, Dr Sam Ellis, Prof Dawn Skelton or if unavailable the chief investigator can facilitate interviews, to ensure a suitably experienced member of the team is involved in supporting an in-depth conversation into participants experience of the study intervention. The chief investigator will ideally not undertake these interviews to minimise researcher bias or observer effects

Data Analysis Descriptive statistics will be used to express baseline and quantitative data (Mean, mode, percentage spread and range). Changes in pre-post assessments will be examined by comparing means of the same group at a different time point using a paired t-test or an equivalent non-parametric test. Intervention effects will be represented by a point estimate (95% confidence interval). Correlations between baseline information and changes in outcome measure scores will be undertake using a pearsons correlation co-efficient test or similar.

Qualitative analysis of semi-structured interview transcripts will be undertaken using thematic analysis to explore patients perceptions of the intervention. Thematic analysis has been used previously in multiple studies and is able to deliver an accessible and theoretically flexible approach to qualitative data analysis (Braun, 2006).

Data analysis will be undertaken by the chief investigator with support from the supervisory team. The chief investigator will use SPSS to complete data analysis of quantitative data, normality testing, mean comparison, descriptive statistics and correlation calculations. Professor Dawn Skelton will act as a quality reviewer for all quantitative data.

Qualitative data will be reviewed in an iterative process using NVivo version 12 with the chief investigator and Dr Fiona Kennedy independently reviewing the raw transcripts to code and eventually create themes that will be discussed at several points to ensure results are accurate, agreed and transparent. Once coding is completed Dr Sam Ellis will review this coding and theming process and where necessary provide a third opinion where disagreements occur and also confirm the accuracy and agreement of coding and final themes.

ELIGIBILITY:
Inclusion Criteria:

* Older adults - at least 65 years of age or older
* Referred to the NHS falls service and identified as 'at risk of a fall' by the NHS falls team - this will be based on the discretion of the referring falls team. NB participants do not need to have experienced a fall to be included.
* Community dwelling - participants need to be living independently, this can include a package of care or family support
* Be able to ambulate independently with a walking aid (10 meters in a straight line)
* have self-reported visual and auditory capacities to follow the exercises
* have the capacity to provide a signed informed-consent statement based on the Six-item screener score with 2 or more wrong answers indicating a high risk of reduced capacity (Callahan et al, 2002, Carpenter et al, 2011).

Exclusion Criteria:

Participants -

* living in a Residential or Care Home
* unable to follow simple instructions or guidance
* who have a medical contraindication for physical activity, participants will be asked to self-declare in line with the Health Commitment Statement (UKACTIVE,2018)
* unable to ambulate independently 10 meters with a walking aid
* with a severe visual and auditory disabilities
* with an unstable cardiovascular disease
* with a neurological disorder that could compromise them from exercising
* with a lower-extremity fracture in the past year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | 5-10 minutes to administer
  Functional Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Skelton, PhD, Study Director — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No